CLINICAL TRIAL: NCT06288269
Title: Factors of Control Hypertension or Non-insulin-dependent Diabetes Mellitus Type 2 on the Severity of Stroke and Survival Rates Within 1 Year in Trat Province.
Brief Title: Factors of Control Hypertension or Type 2 Diabetes on the Severity of Stroke and Survival Rates Within 1 Year in Trat
Status: Completed | Type: Observational
Sponsor: Phrapokklao Hospital,Thailand (Other)
Responsible Party: Principal Investigator, Panuwat Soponlertpong, Deputy Public Health Doctor of Trat Province, Phrapokklao Hospital,Thailand
Other Study IDs: PhrapokklaoHospital
Record Dates: First submitted 2024-02-02; First posted 2024-03-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stroke; Hypertension; Type2diabetes
Keywords: National Institute of Health Stroke Scale
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control of Hypertension or/and Type 2 Diabetic: Control disease of HT Control disease of DM2 Control disease of HT plus DM2
  Interventions: Other: Severity of Stroke and 1 year survival
- Uncontrol of Hypertension or/and Type 2 Diabetic: Uncontrol disease of HT Uncontrol disease of DM2 Uncontrol disease of HT plus DM2
  Interventions: Other: Severity of Stroke and 1 year survival

INTERVENTIONS:
Other: Severity of Stroke and 1 year survival — Evaluated from NIHSS and clinical outcome 1 year survival death

SUMMARY:
The purpose of this study was to study factors for controlling hypertension or type 2 diabetes before stroke diagnosis on the severity level when a stroke occurs, NIHSS, and survival rate after having a stroke in 1 year in Trat Province The research hypothesis was patients with hypertension or type 2 diabetes who are well-controlled Will have a lower NIHSS score than the group whose disease is not well-controlled. and patients with hypertension or type 2 diabetes that is well controlled There will be a higher survival rate for patients diagnosed with cerebrovascular disease within 1 year than those whose disease cannot be controlled.

DETAILED DESCRIPTION:
BACKGROUND: Situation of Non-communicable disease groups. It was the number one health problem in the world. The situation in Thailand from 2017-2022 found an increase in the number of new diagnoses and death cases from stroke patients. For the situation in Trat Province, it was found that the situation of sickness rates tend to be stable. As for the death rate per 100,000 people from stroke, there was a continuous upward trend. Therefore, a research project was organized to study the factors of control disease (hypertension or non-insulin-dependent diabetes mellitus type 2) on the severity of stroke and survival rates within 1 year to be used as information for further patient care.

OBJECTIVES: To study factors that influence the severity of stroke and correlate with survival rates within 1 year in Trat Province.

METHODS: This is a retrospective analytic cohort study. Data was collected using a Case Record Form (CRF) to record information on a total of 291 cases of hypertension and non-insulin-dependent diabetes mellitus type 2 patients who entered the stroke treatment system at Trat Hospital in the year 2022. Data were analyzed by Chi-square statistics to test the relationship of NCD control with the severity of stroke and using Kaplan-Meier Curve test hypotheses for comparing survival rates using Log-rank test statistics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic hypertension or type 2 diabetes with a history of illness of at least 1 year before the stroke.
* Patients had a new stroke for the first time in his life, including an ischemic stroke. hemorrhagic stroke and hemorrhage in the brain
* The patient was confirmed by CT scan
* Thai nationality.

Exclusion Criteria:

* Patients diagnosed with cerebrovascular disease who have a previous history of ischemic or hemorrhagic stroke.
* Patients diagnosed with transient ischemic attack
* Patients who have a history of chronic disease that are at high risk of having a stroke, such as being a pregnant patient, still taking birth control pills.
* There are certain genetic diseases, such as antiphospholipid syndrome
* Patients had previous history of brain aneurysm, extracranial arterial dissection, atrial fibrillation, drug addict use, etc.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample group of people who have had a stroke in fiscal year 2022 of people living in Trat Province. From the medical records center of Trat Hospital that received a diagnosis of stroke and were admitted to the hospital, a total of 729 cases were taken into the study process with criteria for selecting research participants (Inclusion criteria) and criteria. Exclusion criteria resulted in 291 patients who met the aforementioned criteria. There were 244 patients with hypertension as a comorbidity, 129 patients with type 2 diabetes as a comorbidity, and 100 patients with hypertension and type 2 diabetes as a comorbidity.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Stroke severity was assessed using the National Institute of Health Stroke Scale (Clinical Mild NIHSS = 0-4 and Clinical Moderate to severe NIHSS = 5-42) | Results of controlling diabetes and hypertension in the 1-3 year period before having a stroke.
  Patients with new stroke case with different diseases control will have different severity of stroke.
1 year survival death | 1 year after stroke attack
  Patients with new stroke case with different diseases control will have different death rate in 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Panuwat Soponlertpong, Principal Investigator — Trat Provincial Public Health Office
Locations (1):
- Trat Provincial Public Health Office, Trat, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Division of Noncommunicable Diseases DoDC, Ministry of Public Health,. Report on the situation of NCDs, diabetes, and high blood pressure. and related risk factors 2019. Akson Graphic and design Printing and Publishing 2019. 8-9 p.
- [Background] Kogan E, Twyman K, Heap J, Milentijevic D, Lin JH, Alberts M. Assessing stroke severity using electronic health record data: a machine learning approach. BMC Med Inform Decis Mak. 2020 Jan 8;20(1):8. doi: 10.1186/s12911-019-1010-x. PMID 31914991
- [Background] Tziomalos K, Spanou M, Bouziana SD, Papadopoulou M, Giampatzis V, Kostaki S, Dourliou V, Tsopozidi M, Savopoulos C, Hatzitolios AI. Type 2 diabetes is associated with a worse functional outcome of ischemic stroke. World J Diabetes. 2014 Dec 15;5(6):939-44. doi: 10.4239/wjd.v5.i6.939. PMID 25512800
- [Background] Alawneh KZ, Qawasmeh MA, Raffee LA, Al-Mistarehi AH. Ischemic stroke demographics, clinical features and scales and their correlations: an exploratory study from Jordan. Future Sci OA. 2022 Aug 5;8(7):FSO809. doi: 10.2144/fsoa-2022-0017. eCollection 2022 Aug. PMID 36248068
- [Background] Zhang X, Liu Y, Zhang F, Li J, Tong N. Legacy Effect of Intensive Blood Glucose Control on Cardiovascular Outcomes in Patients With Type 2 Diabetes and Very High Risk or Secondary Prevention of Cardiovascular Disease: A Meta-analysis of Randomized Controlled Trials. Clin Ther. 2018 May;40(5):776-788.e3. doi: 10.1016/j.clinthera.2018.03.015. Epub 2018 Apr 12. PMID 29656857
- [Background] Vemmos KN, Tsivgoulis G, Spengos K, Zakopoulos N, Synetos A, Manios E, Konstantopoulou P, Mavrikakis M. U-shaped relationship between mortality and admission blood pressure in patients with acute stroke. J Intern Med. 2004 Feb;255(2):257-65. doi: 10.1046/j.1365-2796.2003.01291.x. PMID 14746563
- [Background] Ntaios G, Egli M, Faouzi M, Michel P. J-shaped association between serum glucose and functional outcome in acute ischemic stroke. Stroke. 2010 Oct;41(10):2366-70. doi: 10.1161/STROKEAHA.110.592170. Epub 2010 Aug 19. PMID 20724712
- [Background] Hu G, Sarti C, Jousilahti P, Peltonen M, Qiao Q, Antikainen R, Tuomilehto J. The impact of history of hypertension and type 2 diabetes at baseline on the incidence of stroke and stroke mortality. Stroke. 2005 Dec;36(12):2538-43. doi: 10.1161/01.STR.0000190894.30964.75. Epub 2005 Nov 10. PMID 16282538
- [Background] Chang WW, Fei SZ, Pan N, Yao YS, Jin YL. Incident Stroke and Its Influencing Factors in Patients With Type 2 Diabetes Mellitus and/or Hypertension: A Prospective Cohort Study. Front Cardiovasc Med. 2022 Feb 9;9:770025. doi: 10.3389/fcvm.2022.770025. eCollection 2022. PMID 35224030
- [Background] Murphy SJ, Werring DJ. Stroke: causes and clinical features. Medicine (Abingdon). 2020 Sep;48(9):561-566. doi: 10.1016/j.mpmed.2020.06.002. Epub 2020 Aug 6. PMID 32837228
- [Background] American Diabetes Association. Standards of Medical Care in Diabetes-2022 Abridged for Primary Care Providers. Clin Diabetes. 2022 Jan;40(1):10-38. doi: 10.2337/cd22-as01. No abstract available. PMID 35221470
- [Background] Kandil H, Soliman A, Alghamdi NS, Jennings JR, El-Baz A. Using Mean Arterial Pressure in Hypertension Diagnosis versus Using Either Systolic or Diastolic Blood Pressure Measurements. Biomedicines. 2023 Mar 10;11(3):849. doi: 10.3390/biomedicines11030849. PMID 36979828
- See also: World Stroke Organization. WSO Global Stroke Fact Sheet 2022 [Internet]. 2022. — https://www.world-stroke.org/news-and-blog/news/wso-global-stroke-fact-sheet-2022